CLINICAL TRIAL: NCT03273283
Title: Prevenció Dels Problemes Relacionats Amb Alcohol a urgències.
Brief Title: Feasibility and Effectiveness of a Specialized Brief Intervention for Hazardous Drinkers in an Emergency Department.
Acronym: PPAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Antoni Gual, Head of the Addiction Unit, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPAU
Record Dates: First submitted 2017-08-31; First posted 2017-09-06 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients received a brief intervention on alcohol use. This brief intervention was a little chat based on motivational techniques to enhance motivation to reduce alcohol use or to initiate treatment. Patients were referred to specialized treatment when indicated.
  Interventions: Behavioral: Brief Intervention
- Control (No Intervention): Informative leaflets regarding alcohol use

INTERVENTIONS:
Behavioral: Brief Intervention — Patient's received a brief intervention on alcohol use based on motivational techniques, and a referral to treatment when indicated.
  Other Names: Referral to treatment
  Arms: Intervention

SUMMARY:
Alcohol use and its consequences represent an important public health problem. As well as alcohol dependence, hazardous drinking also contributes to a high burden in terms of morbidity and mortality. To improve these patients' prognosis and decrease associated social and health care costs, it is necessary to increase early detection, intervention and treatment for these problems. For these reasons, SBIRT programmes (Screening Brief Intervention and Referral to Treatment) have been developed, evaluated and shown to be effective, particularly in primary care and general practice. Nevertheless, effectiveness of SBIRT in emergency departments (ED) has not been clearly established.

The investigators aimed to evaluate the feasibility and efficacy of an SBIRT programme in the ED of a tertiary hospital.

DETAILED DESCRIPTION:
The investigators conducted a randomized controlled trial to study the feasibility and efficacy of an SBIRT programme for hazardous drinkers presenting in an ED. All patients older than 18 years old attending the emergency department were potentially eligible. Cognitively impaired or medically unstable patients were excluded. Patients seeking treatment for alcohol use were also excluded. Patients were randomized to two groups, with the control group receiving two leaflets - one regarding alcohol use, and the other giving information about the study protocol. The intervention group received the same leaflets as well as a brief motivational intervention on alcohol use; and, where appropriate, a referral to specialised treatment. The primary outcomes were the proportion of hazardous drinkers measured by AUDIT-C scale and the proportion of patients attending specialised treatment at 1.5 and 4.5 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 or older attending to the emergency department were potentially eligible patients
* Patients with an AUDIT-C score higher than 6 points for men and 5 for woman were invited to participate

Exclusion Criteria:

* Cognitive impairment
* Medically unstable
* Patients explicitly demanding alcohol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-01 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
There is nno plan, but we have already shared and will continue sharing them
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Since de beginning and for 5 years
Access Criteria: For scientific purposes

REFERENCES:
- [Derived] Bruguera P, Barrio P, Manthey J, Oliveras C, Lopez-Pelayo H, Nuno L, Miquel L, Lopez-Lazcano A, Blithikioti C, Caballeria E, Matrai S, Rehm J, Vieta E, Gual A. Mid and long-term effects of a SBIRT program for at-risk drinkers attending to an emergency department. Follow-up results from a randomized controlled trial. Eur J Emerg Med. 2021 Oct 1;28(5):373-379. doi: 10.1097/MEJ.0000000000000810. PMID 33709997

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 99 | 101
Completed | 72 | 81
Not Completed | 27 | 20

BASELINE CHARACTERISTICS:
Population: At baseline, participants' demographic and enrollment-related characteristics were compared across treatment conditions using t- and chi-square tests according to the nature of each variable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (16.2) | 44 (17.1) | 42.81 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 71 | 73 | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Alcohol related presenting condition [Count of Participants; unit: Participants] — Those patients attended on ED for a condition directly related to their alcohol consumption, such as alcohol intoxications, accidents, liver diseases...
  Participants | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Risky Drinkers Measured by AUDIT-C
Description: We assessed participants with AUDIT-C (a tool to assess alcohol consumption). Main outcome 1 is the proportion of patients who score more than 6 i men and 5 in women in this scale.
  AUDIT-C is the short version of the AUDIT scale (Alcohol use disorders identification test). Consists of a three items scale ( frequency of alcohol consumption, amount of alcohol units per day of consumption and frequency of binge drinking), and ranges from 0 (abstinence) to 12 (very high alcohol use). The higher the score is, the more important the alcohol use is, and more risk of presenting an alcohol use disorder.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 72 | 81
Participants | 20 | 39

2. Primary Outcome: Proportion of Patients Attending to Specialized Treatment
Description: Proportion of patients that initate specialized treatment to reduce alcohol use
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 72 | 82
Participants | 17 | 8

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: no different definition
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 2/99 | 1/101
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/101
Other Adverse Events (participants affected / at risk) | 0/99 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT03273283/Prot_SAP_000.pdf